CLINICAL TRIAL: NCT00863616
Title: Self-Administered High Frequency Chest Wall Oscillation Technique for Mucus Clearance in COPD: An Exploratory Pilot Project Using the SMARTVEST Device
Brief Title: High Frequency Chest Wall Oscillation in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: Electromed, Inc. (Industry)
Responsible Party: Indranil Chakravorty/ Consultant Physician, East & North Herts NHS Trust
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06/Q0303/57
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Mucus hypersecretion; HRQL; ESWT; HFCWO
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HFCWO (Experimental): HFCWO twice a day delivered by SmartVest device at 13Hz FOR 20min x2. Duration 4 weeks in each phase with a 2week washout.
  Interventions: Device: HFCWO - SmartVest
- Placebo/Control (No Intervention): Self-administered breathing exercises

INTERVENTIONS:
Device: HFCWO - SmartVest — SmartVest with vest administered for 20min at 11-13Hz
  Other Names: SmartVest
  Arms: HFCWO

SUMMARY:
Patients with Chronic obstructive pulmonary disease (COPD) tend to have cough, excess mucus production and breathlessness as cardinal features. The excess mucus production often leads to frequent infections, exacerbations and poor quality of life. Mucociliary clearance may have an impact on improving symptoms, exercise tolerance, quality of life and reduce exacerbations.

High frequency chest wall oscillation(HFCWO) devices use percussion to the chest wall delivered from a pump through a close fitting inflatable vest. This technique has been shown to enhance mucus clearance in patients with cystic fibrosis and Bronchiectasis. This pilot study was designed to explore the feasibility, tolerance and effectiveness of the HFCWO in patients with advanced COPD.

DETAILED DESCRIPTION:
1.1 Background

Chronic obstructive pulmonary disease (COPD) is a major health problem across the world and its medical, societal and economic impacts continue to grow. COPD is characterized by chronic obstruction of expiratory flow affecting peripheral airways, associated with chronic bronchitis (mucus hypersecretion with goblet cell and submucosal gland hyperplasia) and emphysema (destruction of airway parenchyma), together with fibrosis and tissue damage, and inflammation of the small airways1. The beneficial effects of smoking cessation in slowing the decline in lung function and the progression of disease have been clearly established. Whether other factors such as mucus hypersecretion, respiratory infections and airway hyper-reactivity contribute to disease progression independent of cigarette smoking is still being debated2.

Patients with COPD are often distressed by mucus hypersecretion which is one of the hallmarks of the disease but little is known about the impact of current therapies on mucus hypersecretion due to the logistical challenges of objectively quantifying mucus in clinical studies 3. Mucus hypersecretion occurs as a direct result of airway inflammation. Neutrophils that die by necrosis disgorge proteases and reactive oxygen species into the lumen. It is concluded that neutrophil death via necrosis leads to the high concentrations of free neutrophil elastase and reactive oxygen species in the sputum of patients with airway neutrophilia and mucus hypersecretion. Inflammatory cells (neutrophils), molecules (neutrophil elastase and reactive oxygen species), signaling pathways (EGFR), and cellular processes (neutrophil necrosis) contribute to mucus hypersecretion in COPD4.

Mucus hypersecretion leads to increased work of breathing, reduced exercise tolerance, deteriorating lung function and increases dyspnoea and cough. Often the mucus hypersecretion also interferes with nocturnal sleep and has a further negative impact on health related quality of life. Combined mucus hypersecretion, reduced clearance, and impairment of the lung defence mechanisms explain why COPD patients even with stable condition, carry potential respiratory pathogens in significant concentration, paving the way for infection and acute exacerbations of COPD5;6. In the natural history of COPD chronic mucus hypersecretion is thought to be linked to the accelerated decline of forced expiratory volume in one second (FEV1)5 7 .

Although mucoactive drugs (which improve the ease of mucus clearance) may be effective in mucus hypersecretion, the uncertainty surrounding their effectiveness, due primarily to the relative lack of evidence from randomised controlled trials and an uncertainty from epidemiological studies linking mucus hypersecretion with mortality8-11, have led to their poor diffusion and adoption in international guidelines 7. However, in combination with newer therapeutic strategies currently in research and development phase targeting airway inflammation and thus reducing mucus hypersecretion, there is a renewed interest in re-evaluating mucus clearance strategies in improving HRQL, exacerbations and morbidity associated with COPD 12;13.

Airway clearance forms a vital part the management of patients with CF14, Bronchiectasis and neuro-muscular diseases15 and has a positive impact on lung function, infection rate and mortality16;17. Individually tailored chest physiotherapy18 with forced expiratory manoeuvres is often considered the gold standard in airway clearance19, although self-administered techniques may be equally effective20 and preferred by patients17;21. Self-administered airway clearance techniques using devices which create a turbulent airflow thus encourage shearing of mucus from bronchial wall, have shown promise in improving HRQL and function in COPD patients22.

High frequency chest wall oscillation (HFCWO)23 is known to reduce respiratory rate but improve ventilation in patients with COPD24 and CF25. Experimental results suggest that shearing at the air-mucus interface could be a significant factor in the enhanced tracheal mucus clearance during HFCWO26. Unlike in CF patients who often have greater support from family members and show high levels of motivation and thus compliance in adhering to self-administered airway clearance techniques, COPD patients have low motivation and poor compliance. Thus self-administered techniques for mucosal clearance may be less effective in clinical settings away from dedicated research programs. Thus the HCFWO may offer a more passive modality of airway clearance with consequently higher compliance, if found to be equally effective and well-tolerated in this group of patients. If HFCWO is shown to improve HRQL, symptoms and exercise tolerance then it may have a significant role in reducing exacerbations and hospital admissions as well as allowing effective management in the community setting. The cost benefit of such improvements will need to be explored in larger studies in the future.

ELIGIBILITY:
Inclusion Criteria:

1. COPD; patients defined by a history of cough, breathlessness and/ mucus/sputum production with lung function showing FEV1/FVC <70% and FEV1<80% predicted and < 20% reversibility from baseline on administration of nebulised b2-agonist (Salbutamol 5mg)
2. Age 40-85 years
3. Mucus hypersecretion ( > 25 ml/72 h collection)

Exclusion Criteria:

1. Chest wall deformity (i.e., kyphoscoliosis, Rib fractures)
2. Severe osteoporosis
3. Haemoptysis within the last 3 months
4. Thoracic or abdominal surgery within 3 months
5. Respiratory failure on non-invasive ventilator therapy
6. Tracheostomy or neck deformities
7. Neuro-muscular dysfunction or disability (i.e., Paralysis due to cerebrovascular disease) which may make it impossible to use the device safely
8. Congestive heart failure (decompensated)
9. Any other mucolytic therapy
10. Significant hiatus hernia or gastro-esophageal reflux disease
11. Recent myocardial infarction or unstable angina

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Health related quality of life (St George's Respiratory Questionnaire) | 3 months

SECONDARY OUTCOMES:
Exercise tolerance (Endurance Shuttle Walk Time achieved) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Indranil Chakravorty, PhD, MRCP, Principal Investigator — East & North Herts NHS Trust, Stevenage, Herts, UK
Locations (1):
- East & North Herts NHS Trust, Stevenage, Herts, United Kingdom

REFERENCES:
- [Derived] Chakravorty I, Chahal K, Austin G. A pilot study of the impact of high-frequency chest wall oscillation in chronic obstructive pulmonary disease patients with mucus hypersecretion. Int J Chron Obstruct Pulmon Dis. 2011;6:693-9. doi: 10.2147/COPD.S22896. Epub 2011 Dec 14. PMID 22259246